CLINICAL TRIAL: NCT01729676
Title: Impact of the Geographical FACTor on the Prostate Cancer Stage at Hormonal Therapy Initiation: FACT STUDY
Brief Title: Impact of the Geographical FACTor on the Prostate Cancer Stage at Hormonal Therapy Initiation
Acronym: FACT
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000059
Record Dates: First submitted 2012-10-23; First posted 2012-11-20 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group A: Degarelix or gonadotrophin releasing hormone (GnRH) agonist for treatment of prostate cancer according to physicians current practice
  Interventions: Drug: Degarelix or GnRH agonist

INTERVENTIONS:
Drug: Degarelix or GnRH agonist — Degarelix or GnRH agonist for treatment of prostate cancer according to physicians current practice

SUMMARY:
French epidemiological data have shown a heterogeneous distribution of the risk of mortality from prostate cancer according to region. The main objective is to describe the distribution of prostate cancer stages when first line hormonal therapy is introduced (overall and by region).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically demonstrated prostatic adenocarcinoma.
* Patients never previously treated with hormonal therapy for prostate cancer.
* Patients eligible for hormonal therapy after initial consultation (alone or in combination with curative treatment).
* Patients agreeing to the collection of personal health data for the purposes of the study.
* Patients with locally advanced or metastatic prostatic cancer tumours or a biological recurrence after curative treatment.

Exclusion Criteria:

* Patients participating in a clinical study involving prostate cancer at the time of inclusion in the investigation.
* Patients having received or currently receiving hormonal treatment for prostate cancer (surgical castration or other hormonal manipulation, including GnRH receptor antagonists, antiandrogens, oestrogens, 5 alpha reductase inhibitors).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men never previously treated with hormononal therapy for prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Estimated percentage of different prostate cancer stages (overall and by region) | During a single consultation when first-line prostate cancer hormone therapy is started
  The stages of prostate cancer are classified as locally advanced, metastatic and biological recurrence.

SECONDARY OUTCOMES:
The characteristics of the patients with prostate cancer by region | During a single consultation when first-line prostate cancer hormone therapy is started
  Characteristics are described by demography, tumour characteristics, Gleason score, D'Amico score, prostate specific antigen (PSA), Testosterone and treatment history
The influence of regional factors on staging of prostate cancer | During a single consultation when first-line prostate cancer hormone therapy is started
  The regional influence will be demonstrated by modelling the probability of a patient being at one of the cancer stages (locally advanced cancer, metastatic cancer, biological recurrence).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Hôpital Robert Boulin, Libourne, France